CLINICAL TRIAL: NCT06710288
Title: A Phase 2, Open-label, Single-arm Study Of Autologous Memory Cytokine Enriched Natural Killer (M-CENK) Adoptive Cell Therapy And N-803 (IL-15 Superagonist) In Combination With Gemcitabine In Participants With Recurrent Platinum-Resistant High-Grade Ovarian Cancer
Brief Title: A Phase 2, Open-label, Single-arm Study Of Autologous M-CENK Adoptive Cell Therapy And N-803 (IL-15 Superagonist) In Combination With Gemcitabine In Participants With Recurrent Platinum-Resistant High-Grade Ovarian Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ResQ209
Record Dates: First submitted 2024-11-05; First posted 2024-11-29 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Platinum-resistant Ovarian Cancer
Keywords: high grade ovarian cancer; M-CENK; N-803
MeSH Terms: interventions — Gemcitabine; ALT-803

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All subjects (Experimental): Gemcitabine plus M-CENK plus N-803
  Interventions: Drug: Gemcitabine; Biological: N-803; Biological: M-CENK

INTERVENTIONS:
Drug: Gemcitabine — Dose: 800 mg/m2 intravenously (IV) Frequency: administered on Day 1, Day 8, and Day 15 of each cycle (every 4 weeks)
  Other Names: gemcitabine hydrocholoride; Gemzar
Biological: N-803 — Dose: fixed dose of 1.2 mg subcutaneously (SC) Frequency: administered on Day 1 and Day 15 of each cycle starting at Cycle 2 (every 4 weeks) and when the last dose of M-CENK is administered, N-803 will be administered on Days 1 and 15 of the same cycle followed by 3 additional doses, 2 weeks apart (total of 5 N-803 doses).
Biological: M-CENK — Dose: 0.15 to 0.75 × 109 cells per infusion intravenously (IV) Frequency: administered on Day 1 of each cycle as long as M-CENK cells are available.
  Other Names: Autologous Memory Cytokine Enriched Natural Killer

SUMMARY:
This is phase 2 single arm study evaluating the safety and preliminary efficacy of M-CENK adoptive cell therapy and fixed dose of N-803 in combination with gemcitabine in participants with platinum-resistant high-grade ovarian cancer (HGOC).Up to 20 participants will receive M-CENK (IV) and N-803 (SC) in combination with gemcitabine (IV).

Participants will undergo an apheresis procedure for the collection of mononuclear cells (MNCs) at least 1 day prior to Cycle 1 for manufacturing of M-CENK. Starting in Cycle 1, participants will receive gemcitabine and starting in Cycle 2 they will also receive M-CENK and N-803, until no additional M-CENK is available or confirmed PD per iRECIST, unless the participant is potentially deriving benefit per Investigator's assessment.

Participants who complete the study treatment or discontinue study treatment will be followed for survival/disease status every 12 weeks (± 2 weeks) for up to 12 months after the last study treatment or until death, lost to follow-up, or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years and <85 years old.
2. Able to understand and provide a signed informed consent that fulfills the relevant Institutional Review Board (IRB) or Independent Ethics Committee (IEC) guidelines.
3. Participants must be appropriate for single-agent therapy as the next line of therapy, as determined by the Investigator.
4. Participants must have received prior treatment with bevacizumab.
5. Confirmed diagnosis of platinum-resistant high-grade epithelial ovarian cancer, primary peritoneal or fallopian tube. Platinum-resistant is defined as a relapse within 6 months of receiving 1 to 3 platinum-based chemotherapy regimens.
6. Must have at least one lesion that meets the definition of measurable disease defined by RECIST v1.1 criteria.
7. Must have received at least one but no more than three prior systemic lines of anticancer therapy and had progressive disease (PD) while receiving or immediately after receiving the previous therapy. Progression will be calculated from the date of the last administered dose of platinum based therapy to the date of radiographic imaging that showed evidence of progression.

   * Participants who had received one line of platinum-based therapy must have received at least four cycles of their initial platinum-containing regimen, had a response (complete or partial), and then had PD between 3 and 6 months after their last dose.
   * Participants who had previously received two or three lines of platinum-based therapy must have had PD while receiving the therapy or within 6 months after the last dose.
8. Participants with germline or somatic BRCA1 or BRCA2 mutations must have received prior PARP inhibitor therapy as maintenance or treatment.
9. Must have adequate peripheral venous access on both arms, or be willing to have temporary vascular access placed for apheresis collection, if deemed necessary by the Investigator.
10. Must be able to sit or recline with limited movement for approximately 6 hours during apheresis procedure.
11. Participants must have been previously tested for FRα. If the test result was positive, they must have been offered treatment with mirvetuximab soravtansine-gynx.
12. Agreement to practice effective contraception for female participants of childbearing potential. Female participants of childbearing potential must agree to use effective contraception for up to 7 months after completion of study treatment. Effective contraception includes surgical sterilization (eg, tubal ligation), orals, injectables, 2 forms of barrier methods (eg, diaphragm), intrauterine devices (IUDs), and hormonal therapy.
13. Eastern cooperative oncology group (ECOG) performance status of ≤ 1.
14. Major surgery must be completed and recovered at least 4 weeks prior to the first dose of study treatment.
15. Participants must meet the following organ and marrow function as defined below:

    * Absolute neutrophil count ≥ 1,000/mm3
    * Platelets ≥ 100,000/mm3
    * AST(SGOT)/ALT(SGPT) ≤ 3 × institutional ULN
    * Total bilirubin ≤1.5 × institutional upper limit of normal (ULN) (except Gilbert's or disease-related hemolysis, then < 3 × ULN)
    * Albumin ≥ 3.0 g/dL
    * Serum creatinine ≤ 2.0 mg/dL OR creatinine clearance ≥ 40 mL/min/1.73 m2 by Cockcroft-Gault Formula (Appendix C.1)
    * Oxygen saturation: ≥ 90% on room air
16. Participants with a prior malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
17. Known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association (NYHA) Functional Classification (Appendix B.2). To be eligible for this trial, participants should be class 2B or better.
18. Expected survival > 16 weeks.
19. Stated willingness to comply with study procedures.
20. Able to attend required study visits and return for adequate follow-up, as required by this protocol.

All inclusion criteria must be answered "yes" for a participant to participate in the trial.

Exclusion Criteria:

In order to participate in the study, participants must not meet any of the following criteria:

1. Participants with clear cell, mucinous, or sarcomatous histology, mixed tumors containing any of the above histologies, or low grade or borderline ovarian tumor.
2. Distant metastasis outside of the abdominopelvic cavity (e.g., central nervous system, pulmonary, osseous, etc.).
3. Have had anti-tumor chemotherapy or other investigational agents within 2 weeks prior to M-CENK cell infusion, or immunotherapy within 4 weeks prior, or those who have not recovered from adverse events due to agents administered more than two weeks prior. The intent of the language is to ensure that anti-tumor chemotherapy or other investigational agents are not administered to participants within the specified window since they can potentially affect M-CENK cell activity. Therefore, the washout period is defined by time from NK cell infusion and not patient enrollment. During eligibility confirmation from the study team is requested to confirm that according to the planned M-CENK cell dosing schedule, the washout period should be completed, based on each drug class.
4. Current bowel obstruction, history of bowel obstruction, or high risk for bowel obstruction (in the opinion of the investigator).
5. Poor oral intake requiring parenteral nutrition or dependence on intravenous fluids.
6. Presence or history of ascites.
7. Receiving any other investigational agents.
8. Solid organ transplant (allograft) recipients.
9. Known additional malignancy that is progressing or requires active treatment, or history of other malignancy within 2 years of the first dose of study treatment with the exception of cured basal cell or squamous cell carcinoma of the skin, superficial bladder cancer, carcinoma in situ of the cervix, or other non-invasive or indolent malignancy, or cancers from which the patient has been disease-free for > 1 year after treatment with curative intent.
10. Known hypersensitivity or anaphylaxis to sulfa-containing study medication(s).
11. Known allergy to dimethyl sulfoxide (DMSO).
12. Prior history of immune-related toxicity during immune therapy that resulted in permanent discontinuation of therapy (as recommended per product label or consensus guidelines) OR any immune-related toxicity requiring intensive or prolonged immunosuppression to manage (with the exception of endocrinopathy that is well-controlled on replacement hormones) are excluded.
13. Autoimmune disease: history of inflammatory bowel disease, including ulcerative colitis and Crohn's disease, are excluded from this study, as are patients with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [Wegener's granulomatosis]) and motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre syndrome and myasthenia gravis). participants with Hashimoto thyroiditis are eligible.
14. Systemic corticosteroid therapy (> 10 mg of prednisone or equivalent dose of systemic steroids for at least 4 weeks prior to NK cell infusion). The intent of this language is to ensure that systemic steroids are not administered to participants within the specified window since this can potentially affect NK cell activity. Therefore, the washout period is defined by time from NK cell infusion and not patient enrollment. During eligibility confirmation the study team is requested to confirm that according to the planned NK cell dosing schedule, the washout period should be completed.
15. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
16. HIV-positive participants are ineligible because of the potential for pharmacokinetic interactions with anti-retroviral agents used in this study. In addition, these participants are at increased risk of lethal infections when treated with marrow-suppressive therapy.
17. Active uncontrolled hepatitis B or C are ineligible as they are at high-risk of lethal treatment-related hepatotoxicity in the setting of marrow suppression. Known non-infectious pneumonitis or any history of interstitial lung disease.
18. Receipt of a live vaccine within 30 days of start of study treatment. During eligibility confirmation the study team is requested to confirm that according to the planned NK cell dosing schedule, the washout period should be completed.

All exclusion criteria must be answered "no" for a participant to participate in the trial.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Evaluate Progression Free Survival (PFS) | Cycle 1 Day 1 through End of Study, up to 2 years
  Measured by RECIST v1.1 and iRECIST
Evaluate Overall Survival (OS) | Cycle 1 Day 1 through End of Study, up to 2 years
Evaluate Objective Response Rate (ORR) | Cycle 1 Day 1 through End of Study, up to 2 years
  Measured by RECIST v1.1 and iRECIST
Evaluate Duration of Response (DOR) | From time of first response to the date of disease progression or death, up to 2 years
  Measured by RECIST v1.1 and iRECIST
Evaluate Disease Control Rate (DCR) | Cycle 1 Day 1 through End of Study, up to 2 years
  Measured by RECIST v1.1 and iRECIST
Evaluate the time to progression or death on the next line of treatment (PFS2) of participants receiving M-CENK adoptive cell therapy and N-803 in combination with gemcitabine. | Cycle 1 Day 1 through End of Study, up to 2 years
  Measured by RECIST v1.1 and iRECIST and survival status
Evaluate the CA-125 response rate (RR) per Gynecologic Cancer Intergroup (GCIC) CA-125 criteria. | Cycle 1 Day 1 through End of Study, up to 2 years
  Measured by the CA-125 result

SECONDARY OUTCOMES:
Safety: Evaluate adverse events | Apheresis to 30 days after the last dose of study treatment or the end of treatment visit, up to 13 months
Safety: Incidence of clinically significant changes in comprehensive metabolic panel (CMP) | Screening through Follow-up, up to 2 years
  Standard blood chemistry panel made up of 14 separate chemistry measurements so can detect a range of abnormalities in blood sugar, nutrient balance, and liver and kidney health. Each clinical site will use their local laboratory upper limit of normal (ULN) range. The treating investigator will assess each result composing the CMP and determine if each result is within expected normal range or outside of the expected normal range.
Safety: Incidence of clinically significant changes in Hematology blood panel | Screening through Follow-up, up to 2 years
  Blood test checking the levels for White Blood Cell, Red Blood Cell, Platelets, Hemoglobin, Hematocrit, Basophils, Eosinophils, Lymphocytes, Monocytes and Neutrophils per unit volume. Each clinical site will use their local laboratory upper limit of normal (ULN) range. The treating investigator will assess each component of the Hematology panel and determine if each result is within expected normal range or outside of the expected normal range.
Safety: Incidence of clinically significant changes in Temperature | Screening through Follow-up, up to 2 years
  Temperature measured in either Fahrenheit or Celsius and for any abnormalities. Each site will assess to determine if temperature is within expected normal range or outside of the expected normal range.
Safety: Incidence of clinically significant changes in Heart Rate | Screening through Follow-up, up to 2 years
  Heart rate measured in beats/minute. Each site will assess to determine if heart rate is within expected normal range or outside of the expected normal range.
Safety: Incidence of clinically significant changes in Respiratory Rate | Screening through Follow-up, up to 2 years
  Respiratory rate measured in breaths/minute. Each site will assess to determine if respiratory rate is within expected normal range or outside of the expected normal range.
Safety: Incidence of clinically significant changes in Blood Pressure | Screening through Follow-up, up to 2 years
  Blood pressure measured in Systolic and Diastolic mmHg. Each site will assess to determine if blood pressure is within expected normal range or outside of the expected normal range.
Safety: Incidence of clinically significant changes in Oxygen Saturation | Screening through Follow-up, up to 2 years
  A pulse oximeter measures oxygen saturation as a percentage. Determines the ratio of the current levels of oxygenated hemoglobin to deoxygenated hemoglobin. Each site will assess to determine if oxygen saturation is within expected normal range or outside of the expected normal range.

OTHER OUTCOMES:
Exploratory: Evaluate the number and phenotype of M-CENK cells performed by flow cytometry and mass cytometry (CyTOF). | During M-CENK production between Apheresis and Cycle 2 Day 1, up to 2 months
Exploratory: Characterize the functionality of M-CENK cells as measured by intracellular staining for cytokines, surface marker staining, and assessments of cytotoxicity. | During M-CENK production between Apheresis and Cycle 2 Day 1, up to 2 months
Exploratory: Assess serum cytokine levels before and after M-CENK infusions. | Cycle 2 Day 1 through last dose of M-CENK, up to 13 months

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Sender, MD, Study Director — ImmunityBio, Inc.
Locations (2):
- United States (2):
  - Chan Soon-Shiong Institute for Medicine, El Segundo, California
  - Hoag, Newport Beach, California